CLINICAL TRIAL: NCT02125604
Title: A Multicenter, Open-Label, Single-Arm Study to Evaluate Gastrointestinal Tolerability in Subjects With Relapsing-Remitting Multiple Sclerosis Receiving Dimethyl Fumarate (TOLERATE)
Brief Title: Gastrointestinal Tolerability Study Of Dimethyl Fumarate In Participants With Relapsing-Remitting Multiple Sclerosis In Germany
Acronym: TOLERATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS407; 2013-001486-17 (EudraCT Number)
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Gastrointestinal event
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dimethyl Fumarate (Experimental): Dimethyl fumarate administered orally at 120 mg twice daily (BID) for the first 7 days and 240 mg BID thereafter for a total of 12 weeks.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — capsules administered according to the prevailing product label
  Other Names: BG00012; Tecfidera; DMF

SUMMARY:
The primary objective of this study is to evaluate the effect of symptomatic therapies on gastrointestinal-related events reported by participants with relapsing-remitting multiple sclerosis initiating therapy with BG00012 (dimethyl fumarate, DMF) in the clinical practice setting.

The secondary objectives of this study in this study population are as follows: to evaluate gastrointestinal-related events requiring symptomatic therapy and the role of those therapies over time; to evaluate gastrointestinal-related events that lead to a physician's decision to manage the events with BG00012 dose modification; and to evaluate gastrointestinal-related events that lead to BG00012 discontinuation after the use of symptomatic therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a confirmed diagnosis of relapsing-remitting multiple sclerosis according to the current McDonald Criteria and satisfy the therapeutic indication as described in the official local registration for Tecfidera (dimethyl fumarate)
* Naïve to dimethyl fumarate and fumaric acid esters

Key Exclusion Criteria:

* Female subjects who are currently pregnant or breastfeeding or who are considering becoming pregnant while in the study
* History of significant gastrointestinal disease (e.g., irritable bowel disease, peptic ulcer disease, history of major gastrointestinal surgeries), or chronic use of gastrointestinal-related symptomatic therapy as determined by the Investigator (or ≥ 7 consecutive days of gastrointestinal-related symptomatic therapy
* Known active malignancies
* History of anaphylaxis or severe allergic reactions or known drug hypersensitivity
* Current use of B vitamin supplements
* In the opinion of the Investigator, blood test values suggestive of a low lymphocyte count or renal or hepatic impairment, as described in the product label precautions for use

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (19):
- Germany (19):
  - Research Site, Augsburg
  - Research Site, Bamburg
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Erbach im Odenwald
  - Research Site, Erlangen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, Minden
  - Research Site, Mittweida
  - Research Site, München
  - Research Site, Münster
  - Research Site, Osnabrück
  - Research Site, Potsdam
  - Research Site, Siegen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 214 participants were screened and enrolled; 3 participants did not receive study drug (1 withdrew consent and 2 did not meet all inclusion/exclusion criteria). A total of 211 participants were included in the safety population.
Groups:
- Dimethyl Fumarate: Dimethyl fumarate administered orally at 120 mg BID for the first 7 days and 240 mg BID thereafter for a total of 12 weeks.
Period: Overall Study
Arm/Group | Dimethyl Fumarate
Started | 211 (enrolled and received at least 1 dose of study drug)
Completed | 180
Not Completed | 31
Not completed — Other | 4
Not completed — Investigator Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Consent Withdrawn | 4
Not completed — Adverse Event | 20

BASELINE CHARACTERISTICS:
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.09 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Utilized Symptomatic Therapy With Gastrointestinal-Related Events During the 12-Week Treatment Period: Modified Overall Gastrointestinal Symptom Scale (MOGISS)
Description: The MOGISS is a questionnaire about the severity of overall gastrointestinal-related events, including specifically symptoms of nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, indigestion, constipation, bloating, and flatulence for 24 hours before the AM dose. Participants who rated the intensity of symptoms reported on the MOGISS and included each symptomatic therapy used in the eDiary are presented.
Time Frame: Up to Week 12
Population: Safety Population: all participants who received at least 1 dose of dimethyl fumarate; n=participants with an assessment during given time period.
Measure: Number; unit: Participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 211
Participants
  Overall Treatment Period; n=211 | 82
  Weeks 1-4; n=211 | 71
  Weeks 5-8; n=186 | 33
  Weeks 9-12; n=178 | 22

2. Primary Outcome: Number of Participants Who Utilized Symptomatic Therapy With Gastrointestinal-Related Events During the 12-Week Treatment Period: Modified Acute Gastrointestinal Symptom Scale (MAGISS)
Description: The MAGISS is a questionnaire in which participants reported overall acute gastrointestinal-related events, (especially symptoms of nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, indigestion, constipation, bloating, and flatulence) for each 10 hours after the AM and PM doses of study drug. Participants who rated the intensity of gastrointestinal-related events reported on MAGISS, included the duration of the gastrointestinal-related events and each symptomatic therapy used in the eDiary are presented.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 211
Participants
  Overall Treatment Period; n=211 | 83
  Weeks 1-4; n=211 | 72
  Weeks 5-8; n=189 | 34
  Weeks 9-12; n=180 | 26

3. Primary Outcome: Worst Severity Of Gastrointestinal-Related Events In Participants Who Utilized Symptomatic Therapy During the 12-Week Treatment Period, MOGISS
Description: The MOGISS is a questionnaire about overall events related to the gastrointestinal system (including nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, indigestion, constipation, bloating, and flatulence) during the 24 hours prior to each AM dose. MOGISS is based on a 0- to 10-point scale, with 0 representing absence of symptoms and 10 representing the most severe symptoms. The worst overall severity score for gastrointestinal-related events was calculated for each participant for the overall treatment period of 12 weeks, and for each 4-week period therein.
Time Frame: Up to Week 12
Population: Safety Population: all participants who received at least 1 dose of dimethyl fumarate and used symptomatic therapy; n=participants with an evaluable assessment during given time period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 84
units on a scale
  Overall treatment period; n=84 | 5.94 (2.427)
  Week 1-4; n=73 | 5.75 (2.554)
  Week 5-8; n=38 | 3.53 (2.533)
  Week 9-12; n=29 | 3.1 (2.568)

4. Primary Outcome: Worst Severity Of Gastrointestinal-Related Events In Participants Who Utilized Symptomatic Therapy During the 12-Week Treatment Period, MAGISS
Description: The MAGISS is a questionnaire about the overall events related to the gastrointestinal system (including nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, indigestion, constipation, bloating, and flatulence) following drug administration (acute symptoms). MAGISS is based on a 0- to 10-point scale, with 0 representing absence of symptoms and 10 representing the most severe symptoms. The worst overall severity score for gastrointestinal-related events was calculated for each participant for the overall treatment period of 12 weeks, and for each 4-week period therein.
Time Frame: Up to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 84
units on a scale
  Overall treatment period; n=84 | 5.93 (2.516)
  Week 1-4; n=73 | 5.88 (2.614)
  Week 5-8; n=39 | 3.31 (2.307)
  Week 9-12; n=29 | 3.55 (2.772)

5. Primary Outcome: Duration of Gastrointestinal-Related Events in Participants Who Utilized Symptomatic Therapy During the 12-Week Treatment Period, MOGISS
Description: The percentage of days with GI events as reported on MOGISS was calculated for each participant and each analysis period using the following formula: 100 x (# of days with [GI] events / # of days tolerability scale completed). The symptomatic therapy (ST) categories were provided by Biogen Medical team as follows: ST1=anti-acid production; ST2=anti-bloating/anti-constipation agent; ST3=multitarget/ herbal agents; ST4=anti-diarrheal (anti-peristaltic); ST5=analgesic (NSAID); ST6=anti-emetic (central); ST7=anti-emetic (pro-kinetic); ST8=antacid; ST9=other; ST10=laxative (pro-kinetic). Overall GI events were reported in the second day after the dose. Relative day for Overall GI events = assessment date-first dose date.
Time Frame: Up to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 84
percentage of days
  Overall treatment period; Any ST (n=84) | 38.13 (29.263)
  Overall treatment period; ST1 (n=50) | 42.08 (27.495)
  Overall treatment period; ST2 (n=26) | 36.98 (29.754)
  Overall treatment period; ST3 (n=20) | 39.61 (29.197)
  Overall treatment period; ST4 (n=16) | 48.15 (30.140)
  Overall treatment period; ST5 (n=10) | 45.94 (27.147)
  Overall treatment period; ST6 (n=8) | 44.33 (29.095)
  Overall treatment period; ST7 (n=6) | 57.52 (21.998)
  Overall treatment period; ST8 (n=5) | 52.71 (31.829)
  Overall treatment period; ST9 (n=3) | 32.78 (26.995)
  Overall treatment period; ST10 (n=2) | 9.20 (2.137)
  Week 1-4; Any ST (n=73) | 49.58 (29.547)
  Week 1-4; ST1 (n=44) | 53.92 (27.197)
  Week 1-4; ST2 (n=23) | 49.53 (32.012)
  Week 1-4; ST3 (n=18) | 55.31 (29.869)
  Week 1-4; ST4 (n=13) | 56.63 (25.764)
  Week 1-4; ST5 (n=9) | 44.42 (32.470)
  Week 1-4; ST6 (n=6) | 48.48 (35.539)
  Week 1-4; ST7 (n=6) | 69.78 (24.808)
  Week 1-4; ST8 (n=5) | 66.43 (31.400)
  Week 1-4; ST9 (n=3) | 41.41 (34.085)
  Week 1-4; ST10 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 5-8; Any ST (n=38) | 41.55 (38.612)
  Week 5-8; ST1 (n=23) | 44.04 (41.414)
  Week 5-8; ST2 (n=3) | 41.67 (52.042)
  Week 5-8; ST3 (n=8) | 37.45 (37.388)
  Week 5-8; ST4 (n=3) | 69.14 (44.186)
  Week 5-8; ST5 (n=3) | 63.75 (31.332)
  Week 5-8; ST6 (n=3) | 70.42 (25.699)
  Week 5-8; ST7 (n=1) | 35.71 (NA) — 1 participant used this symptomatic therapy in this time period.
  Week 5-8; ST8 (n=2) | 56.88 (40.032)
  Week 5-8; ST9 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 5-8; ST10 (n=2) | 1.79 (2.525)
  Week 9-12; Any ST (n=29) | 43.27 (42.322)
  Week 9-12; ST1 (n=15) | 47.66 (43.191)
  Week 9-12; ST2 (n=3) | 82.72 (29.937)
  Week 9-12; ST3 (n=6) | 48.85 (50.931)
  Week 9-12; ST4 (n=4) | 22.12 (20.834)
  Week 9-12; ST5 (n=2) | 62.50 (53.033)
  Week 9-12; ST6 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 9-12; ST7 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 9-12; ST8 (n=2) | 9.26 (13.095)
  Week 9-12; ST9 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 9-12; ST10 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.

6. Secondary Outcome: Percentage of Participants Who First Took Symptomatic Therapy for Gastrointestinal-Related Events at Weeks 4, 8, and 12
Description: The cumulative percentage of dimethyl fumarate-treated participants with relapsing-remitting multiple sclerosis who required symptomatic therapy up to Week 4, Week 8, and Week 12 were estimated using the Kaplan-Meier method.
Time Frame: Week 4, Week 8, Week 12
Population: Safety Population: all participants who received at least 1 dose of dimethyl fumarate and used symptomatic therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 84
percentage of participants
  Week 4 | 35.3
  Week 8 | 38.4
  Week 12 | 41.1

7. Secondary Outcome: Number of Participants Who Used Symptomatic Therapies for Gastrointestinal-Related Events During the 12-Week Treatment Period, by Category
Description: Symptomatic therapies were classified into 10 main categories: anti-acid production (eg, pantoprazole, omeprazole, esomeprazole, ranitidine); anti-bloating/anti-constipation agents (eg, hyoscine butylbromide, sodium picosulfate, Agiolax, dimeticone, lactulose, Movicol, simethicone); multitarget/herbal agents (includes Iberogast, Gaviscon, amaratropfen, Wikalin, Gaviscon & Iberogast, Iberogast & Wikalin); anti-diarrheal (anti-peristaltic; loperamide, racecadotril); analgesic (non-steroidal anti-inflammatory drug [NSAID]; ibuprofen, paracetamol, metamizole); anti-emetic (central; dimenhydrinate, domperidone); anti-emetic (pro-kinetic; metoclopramide); anti-acid (calcium carbonate, magaldrate, sodium hydrogen carbonate, sodium hydroxide/aluminium oxide, Talcid); other (Saccharomyces boulardii, carbon tablet, Lactobacillus acidophilus); laxative (pro-kinetic; bisacodyl). Participants may have taken > 1 symptomatic therapy but were counted only once for the 'All therapies' summary.
Time Frame: Up to Week 12
Population: Safety Population: all participants who received at least 1 dose of dimethyl fumarate and used symptomatic therapy.
Measure: Number; unit: participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 211
participants
  Overall treatment period (OTP): All therapies | 84
  OTP: Anti-acid production | 50
  OTP: Anti-bloating/anti-constipation agent | 26
  OTP: Multi-target/herbal agents | 20
  OTP: Anti-diarrheal (anti-peristaltic) | 16
  OTP: Analgesic (NSAID) | 10
  OTP: Anti-emetic (central) | 8
  OTP: Anti-emetic (pro-kinetic) | 6
  OTP: Antacid | 5
  OTP: Other | 3
  OTP: Laxative (pro-kinetic) | 2
  Week 1-4: All therapies | 73
  Week 1-4: Anti-acid production | 44
  Week 1-4: Anti-bloating/anti-constipation agent | 23
  Week 1-4: Multi-target/herbal agents | 18
  Week 1-4: Anti-diarrheal (anti-peristaltic) | 13
  Week 1-4: Analgesic (NSAID) | 9
  Week 1-4: Anti-emetic (central) | 6
  Week 1-4: Anti-emetic (pro-kinetic) | 6
  Week 1-4: Antacid | 5
  Week 1-4: Other | 3
  Week 5-8: All therapies | 38
  Week 5-8: Anti-acid production | 23
  Week 5-8: Multi-target/herbal agents | 8
  Week 5-8: Analgesic (NSAID) | 3
  Week 5-8: Anti-bloating/anti-constipation agent | 3
  Week 5-8: Anti-diarrheal (anti-peristaltic) | 3
  Week 5-8: Anti-emetic (central) | 3
  Week 5-8: Antacid | 2
  Week 5-8: Laxative (pro-kinetic) | 2
  Week 5-8: Anti-emetic (pro-kinetic) | 1
  Week 9-12: All therapies | 29
  Week 9-12: Anti-acid production | 15
  Week 9-12: Multi-target/herbal agents | 6
  Week 9-12: Anti-diarrheal (anti-peristaltic) | 4
  Week 9-12: Anti-bloating.anti-constipation agent | 3
  Week 9-12: Analgesic (NSAID) | 2
  Week 9-12: Antacid | 2

8. Secondary Outcome: Duration of Use of Symptomatic Therapies for Gastrointestinal-Related Events During the 12-Week Treatment Period, by Category
Description: Symptomatic therapies were classified into 10 categories: anti-acid production (eg, pantoprazole, omeprazole, esomeprazole, ranitidine); anti-bloating/anti-constipation agents (eg, hyoscine butylbromide, sodium picosulfate, Agiolax, dimeticone, lactulose, Movicol, simethicone); multitarget/herbal agents (eg, Iberogast, Gaviscon, amaratropfen, Wikalin, Gaviscon & Iberogast, Iberogast & Wikalin); anti-diarrheal (anti-peristaltic; loperamide, racecadotril); analgesic (NSAID; ibuprofen, paracetamol, metamizole); anti-emetic (central; dimenhydrinate, domperidone); anti-emetic (pro-kinetic; metoclopramide); anti-acid (calcium carbonate, magaldrate, sodium hydrogen carbonate, sodium hydroxide/aluminium oxide, Talcid); other (Saccharomyces boulardii, carbon tablet, Lactobacillus acidophilus); laxative (pro-kinetic; bisacodyl). If a participant had multiple different therapies on the same day, the days on symptomatic therapy was calculated as 1 day in 'All therapies'.
Time Frame: Up to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 84
days
  OTP: All therapies; n=84 | 13.15 (19.21)
  OTP: Anti-acid production; n=50 | 16.62 (22.21)
  OTP: Anti-bloating/anti-constipation agent; n=26 | 2.42 (1.81)
  OTP: Multi-target/herbal agents; n=20 | 9.40 (13.95)
  OTP: Anti-diarrheal (anti-peristaltic); n=16 | 3.13 (2.53)
  OTP: Analgesic (NSAID); n=10 | 3.10 (1.73)
  OTP: Anti-emetic (central); n=8 | 3.25 (4.43)
  OTP: Anti-emetic (pro-kinetic); n=6 | 1.83 (0.98)
  OTP: Antacid; n=5 | 3.60 (4.22)
  OTP: Other; n=3 | 1.67 (0.58)
  OTP: Laxative (pro-kinetic); n=2 | 1.00 (0.00)
  Week 1-4: All therapies; n=73 | 6.03 (6.12)
  Week 1-4: Anti-acid production; n=44 | 7.07 (6.73)
  Week 1-4: Anti-bloating/anti-constipation; n=23 | 2.30 (1.89)
  Week 1-4: Multi-target/herbal agents; n=18 | 3.78 (3.06)
  Week 1-4: Anti-diarrheal (anti-peristaltic); n=13 | 2.62 (1.45)
  Week 1-4: Analgesic (NSAID); n=9 | 2.11 (0.93)
  Week 1-4: Anti-emetic (central); n=6 | 3.17 (3.92)
  Week 1-4: Anti-emetic (pro-kinetic); n=6 | 1.67 (0.82)
  Week 1-4: Antacid; n=5 | 1.80 (1.30)
  Week 1-4: Other; n=3 | 1.67 (0.58)
  Week 5-8: All therapies; n=38 | 10.08 (10.56)
  Week 5-8: Anti-acid production; n=23 | 13.00 (11.14)
  Week 5-8: Multi-target/herbal agents; n=8 | 8.50 (10.45)
  Week 5-8: Analgesic (NSAID); n=3 | 2.00 (1.00)
  Week 5-8: Anti-bloating/anti-constipation; n=3 | 1.33 (0.58)
  Week 5-8: Anti-diarrheal (anti-peristaltic); n=3 | 4.00 (3.61)
  Week 5-8: Anti-emetic (central); n=3 | 2.33 (1.15)
  Week 5-8: Antacid; n=2 | 2.50 (2.12)
  Week 5-8: Laxative (pro-kinetic); n=2 | 1.00 (0.00)
  Week 5-8: Anti-emetic (prokinetic); n=1 | 1.00 (NA) — One participant only was included.
  Week 9-12: All therapies; n=29 | 9.72 (10.31)
  Week 9-12: Anti-acid production; n=15 | 14.73 (10.91)
  Week 9-12: Multi-target/herbal agents; n=6 | 8.67 (8.57)
  Week 9-12: Anti-diarrheal (anti-peristaltic); n=4 | 1.00 (0.00)
  Week 9-12: Anti-bloating/anti-constipation; n=3 | 2.00 (1.00)
  Week 9-12: Analgesic (NSAID); n=2 | 3.00 (0.00)
  Week 9-12: Antacid; n=2 | 2.00 (1.41)

9. Secondary Outcome: Percentage of Participants Who Required Dimethyl Fumarate Dose Reduction In Response To Gastrointestinal-Related Events
Description: Dose reductions are defined as participants who take any dimethyl fumarate 120 mg or 0 mg since initiation of dimethyl fumarate 240 mg.
Time Frame: Up to Week 12
Population: Safety Population: all participants who received at least 1 dose of dimethyl fumarate.
Measure: Number; unit: percentage of participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 211
percentage of participants | 34.6

10. Secondary Outcome: Percentage of Participants Who Discontinued Dimethyl Fumarate Due To Gastrointestinal-Related Treatment-Emergent Adverse Events
Time Frame: Up to Week 12
Population: Safety Population: all participants who received at least 1 dose of dimethyl fumarate.
Measure: Number; unit: percentage of participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 211
percentage of participants | 6.6

11. Primary Outcome: Duration of Gastrointestinal-Related Events in Participants Who Utilize Symptomatic Therapy During the 12-Week Treatment Period, MAGISS
Description: Percentage of days with GI events as reported on MAGISS was calculated for each participant and each analysis period using the following formula: 100 x (# of days with [GI] events / # of days tolerability scale completed). The ST categories were provided by Biogen Medical team as follows: ST1=anti-acid production; ST2=anti-bloating/anti-constipation agent; ST3=multitarget/ herbal agents; ST4=anti-diarrheal (anti-peristaltic); ST5=analgesic (NSAID); ST6=anti-emetic (central); ST7=anti-emetic (pro-kinetic); ST8=antacid; ST9=other; ST10=laxative (pro-kinetic). Overall GI events were reported in the second day after the dose. Relative day for Overall GI events = assessment date-first dose date.
Time Frame: Up to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 84
percentage of days
  Overall treatment period; Any ST (n=84) | 38.20 (30.516)
  Overall treatment period; ST1 (n=50) | 41.29 (29.517)
  Overall treatment period; ST2 (n=26) | 33.67 (27.310)
  Overall treatment period; ST3 (n=20) | 39.28 (29.165)
  Overall treatment period; ST4 (n=16) | 49.94 (33.291)
  Overall treatment period; ST5 (n=10) | 45.65 (27.118)
  Overall treatment period; ST6 (n=8) | 44.71 (30.374)
  Overall treatment period; ST7 (n=6) | 55.32 (23.097)
  Overall treatment period; ST8 (n=5) | 53.42 (31.443)
  Overall treatment period; ST9 (n=3) | 36.92 (27.800)
  Overall treatment period; ST10 (n=2) | 10.88 (1.924)
  Week 1-4; Any ST (n=73) | 51.03 (30.360)
  Week 1-4; ST1 (n=44) | 54.41 (29.608)
  Week 1-4; ST2 (n=23) | 47.84 (30.764)
  Week 1-4; ST3 (n=18) | 56.67 (30.711)
  Week 1-4; ST4 (n=13) | 58.90 (27.111)
  Week 1-4; ST5 (n=9) | 53.74 (32.304)
  Week 1-4; ST6 (n=6) | 46.43 (33.221)
  Week 1-4; ST7 (n=6) | 67.54 (25.296)
  Week 1-4; ST8 (n=5) | 69.86 (28.919)
  Week 1-4; ST9 (n=3) | 47.61 (47.61)
  Week 1-4; ST10 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 5-8; Any ST (n=38) | 40.59 (37.836)
  Week 5-8; ST1 (n=23) | 41.59 (41.442)
  Week 5-8; ST2 (n=3) | 47.14 (45.781)
  Week 5-8; ST3 (n=8) | 38.50 (35.493)
  Week 5-8; ST4 (n=3) | 62.58 (45.775)
  Week 5-8; ST5 (n=3) | 56.33 (33.011)
  Week 5-8; ST6 (n=3) | 71.61 (24.587)
  Week 5-8; ST7 (n=1) | 35.71 (NA) — 1 participant used this symptomatic therapy in this time period.
  Week 5-8; ST8 (n=2) | 62.24 (32.456)
  Week 5-8; ST9 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 5-8; ST10 (n=2) | 10.00 (14.142)
  Week 9-12; Any ST (n=29) | 41.28 (42.466)
  Week 9-12; ST1 (n=15) | 44.24 (44.754)
  Week 9-12; ST2 (n=3) | 76.19 (41.239)
  Week 9-12; ST3 (n=6) | 51.99 (50.113)
  Week 9-12; ST4 (n=4) | 15.48 (10.178)
  Week 9-12; ST5 (n=2) | 63.16 (52.103)
  Week 9-12; ST6 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 9-12; ST7 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 9-12; ST8 (n=2) | 13.11 (7.655)
  Week 9-12; ST9 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.
  Week 9-12; ST10 (n=0) | NA (NA) — No participants used this symptomatic therapy in this time period.

ADVERSE EVENTS:
Time Frame: Serious adverse events: from signing of informed consent through last dose (up to 12 weeks (±5 days) plus 2 weeks (±5 days) follow up. Adverse events: from time of first dose of dimethyl fumarate through last dose (up to 12 weeks (±5 days).
Arm/Group | Dimethyl Fumarate
Serious Adverse Events (participants affected / at risk) | 5/211
Other Adverse Events (participants affected / at risk) | 129/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimethyl Fumarate (N=211)
Multiple sclerosis relapse (Nervous system disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Alanine aminotransferase increrased (Investigations) | 1
Aspartate aminotransferase (Investigations) | 1
Gamma-glutamyltransferase (Investigations) | 1
Alcohol abuse (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dimethyl Fumarate (N=211)
Flushing (Vascular disorders) | 105
Nasopharyngitis (Infections and infestations) | 31
Headache (Nervous system disorders) | 14
Fatigue (General disorders) | 12
Pruritis (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.